CLINICAL TRIAL: NCT04013659
Title: Effect of Gel Renewal During In-office Dental Bleaching Using Violet LED Light as Photo-accelerator. A Randomized Blind Clinical Trial
Brief Title: Effect of Gel Renewal During In-office Dental Bleaching
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Ibirapuera (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Karen Müller Ramalho, Full Professor, Universidade Ibirapuera
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 90670218.3.0000.5597
Record Dates: First submitted 2019-06-09; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Tooth Bleaching

STUDY DESIGN:
Intervention Model Description: Split-mouth model design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G1 - Permanence of the Whitening Gel (Experimental): Permanence of the Whitening Gel (Biological Product: 35% Hydrogen Peroxide) on the tooth enamel during the 15 minutes of dental-bleaching
  Interventions: Other: Dental Bleaching with 35% hydrogen peroxide gel + Violet LED Irradiation
- G2 - Renewal of the Whitening Gel (Experimental): 3 Whitening Gel (Biological Product: 35% Hydrogen Peroxide) renewal every 5 minutes during the 15 minutes of dental-bleaching
  Interventions: Other: Dental Bleaching with 35% hydrogen peroxide gel + Violet LED Irradiation

INTERVENTIONS:
Other: Dental Bleaching with 35% hydrogen peroxide gel + Violet LED Irradiation — After gum protection, the bleaching gel (35% hydrogen peroxide) was applied to the surface of the tooth and irradiated with VIOLET LED

SUMMARY:
Considering the lack of studies related to the violet LED light (405-410nm), applied to tooth whitening, as well as the lack of protocols for its use, this study aims to evaluate if bleaching gel renewal during dental office whitening associated with Violet LED light interferes with final color result and postoperative sensitivity in a randomized, blinded, split-mouth study. Thirty-three volunteers will be selected to participate in the study (n = 33), and the study groups will be: G1 (Permanence of the Whitening Gel on the tooth enamel for 15 minutes) and G2 (3 Whitening Gel renewal every 5 minutes - Total of 15 minutes). In both G1 and G2, teeth will be illuminated with the Violet LED (405-410nm). In the same patient the two treatments (G1 and G2) will be performed, with a split-mouth protocol. The primary outcome will be immediate and mediated color change, quantitatively assessed by colorimetric (color scale) and spectrophotometry tests. Dental sensitivity will also be evaluated during and after tooth whitening using the VAS pain scale. There will be 3 whitening sessions with a 7-day interval between them. The alteration of color and presence of sensitivity will also be evaluated at the times of 14 days and 2 months after the whitening ends. A gel containing 35% hydrogen peroxide will be used. The final color evaluator and responsible for interviewing the patient about the sensitivity will be blind as to which treatment was applied on each side of the patient's arcade.

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene conditions
* Good general health conditions and without systemic disease
* Presence of all teeth, without caries, periodontal disease, restorations, endodontic treatment, crowns
* Patients with dental color A3 or darker, according to the VITA * Classical Color Scale.

Exclusion Criteria:

* Pregnant and lactating female patients
* Presence of caries, periodontal disease or any other infectious source in the oral cavity
* Systematic use of tobacco and alcoholic beverages
* Chronic use of corticosteroids, as well as who makes use of analgesics or anti-inflammatories before or during 48 hours after dental bleaching
* Patients with dentin hypersensitivity
* Patients with tooth color alteration by tetracycline, fluorosis, endodontic treatment.
* Volunteers who use removable prostheses

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Teeth Color 1 | Immediately after treatment
  assessed quantitatively by colorimetric color scale
Teeth Color 2 | Immediately after treatment
  assessed quantitatively by spectrophotometry
Teeth Color 1 | 14 days after treatment
  assessed quantitatively by colorimetric color scale
Teeth Color 2 | 14 days after treatment
  assessed quantitatively by spectrophotometry
Teeth Color 1 | 2 months after treatment
  assessed quantitatively by colorimetric color scale
Teeth Color 2 | 2 months after treatment
  assessed quantitatively by spectrophotometry

SECONDARY OUTCOMES:
Dental sensitivity | Immediately after treatment
  Evaluated through a Visual Analogic Scale (0-10cm) from 0 (no pain) to 10 (maximum pain)
Dental sensitivity | 14 days after treatment
  Evaluated through a Visual Analogic Scale (0-10cm) from 0 (no pain) to 10 (maximum pain)
Dental sensitivity | 2 months after treatment
  Evaluated through a Visual Analogic Scale (0-10cm) from 0 (no pain) to 10 (maximum pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Ibirapuera, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No